CLINICAL TRIAL: NCT04521829
Title: WALKING WITH VIRTUAL REALITY: How Does Optic Flow Speed and Level of Immersion Influence the Gait Pattern in People Post-stroke?
Brief Title: The Effect of Optic Flow Speed Manipulation and the Level of Immersion on the Gait Pattern in People Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University Ghent (Other); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Emma De Keersmaecker, Principal Investigator, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR study - GRAIL/HMD
Record Dates: First submitted 2020-08-03; First posted 2020-08-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: virtual reality; gait; optic flow
MeSH Terms: conditions — Stroke | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-enhanced treadmill walking (Experimental): Participants will be tested during 2 sessions of VR-enhanced treadmill walking.
  Interventions: Other: Walking with different optic flow speeds with 2 different VR devices

INTERVENTIONS:
Other: Walking with different optic flow speeds with 2 different VR devices — Participants will perform 2 sessions of VR-enhanced treadmill walking. One session with the GRAIL system (semi-immersive) and the other session with a fully immersive head-mounted display (Oculus Rift S). In both sessions, the speed of the optic flow will be manipulated: equal to, 2 times faster and 2 times slower than the participant's comfortable walking speed.

SUMMARY:
The aim of this study is to investigate the effect of manipulating the optic flow speed in the virtual environment on the gait pattern during virtual reality (VR) - enhanced treadmill walking in people post-stroke. Furthermore, the study will also investigate if the level of immersion has an effect on the rehabilitation outcomes by manipulating the optic flow speed in two different VR devices: the semi-immersive GRAIL system and the fully-immersive 'Oculus Rift S' HMD.

To properly understand the results of the people with a stroke, we will also investigate the effect of manipulating the optic flow speed and the level of immersion on the gait pattern in healthy people. That way, we can investigate whether virtual reality has a different influence on the gait pattern of people with a stroke than in healthy people.

DETAILED DESCRIPTION:
STUDY DESIGN

This study is an experimental, 2-group, multicenter trial in which people post-stroke and healthy people will perform 2 different sessions of treadmill walking. The 2 sessions will be carried out on 2 separate days within 10 days. Both sessions will be identical, only the VR system used to manipulate the optic flow speed will differ. The order of the 2 sessions and the optic flow speed manipulation will be randomized.

MATERIALS

GRAIL system: The Gait Real-time Interactive Lab (GRAIL) is an integrative motion capture system consisting of 10 optical motion cameras (Vicon Inc., Oxford, UK), a dual belt treadmill with integrated force plates, a 180-degree cylindrical projection screen system, and D-Flow software (Motekforce Link, Amsterdam, Netherlands). The treadmill of the GRAIL system has two modes: fixed walking speed or self-paced. For this study, the treadmill will be self-paced, meaning that the patient is in control and can choose the walking speed. The treadmill will follow the walking speed of the patient, which allow the patient to start, stop and change speed at will. The projection screen of the GRAIL system will assure a semi-immersive virtual environment. The GRAIL system is located in the Smart Space lab (UZ Gent) and will be made available at the researchers of the VUB/UZ Brussel.

Head-mounted display (HMD): The HMD VR system 'Oculus Rift S' (Oculus, LLS, US) is a low-cost HMD that fully integrates the user into the virtual environment by blocking out perception of the real-world. The "Oculus Rift S" will assure a fully immersive virtual environment. The researchers of the VUB/UZ Brussel have the HMD 'Oculus Rift S' in their possession and will make it available for the study.

PROCEDURE

Both sessions will be carried out in the Smart Space lab at the University Hospital of Ghent (Corneel Heymanslaan 10, 9000 Gent) where the GRAIL system is located.

Prior to the start of both sessions, some preparations will have to be done with regard to the outcome measures:

* Patients will be asked to fill in a questionnaire (the Simulator Sickness Questionnaire-Pre).
* Surface electrodes will be placed bilateral on the M. rectus femoris, M. vastus lateralis, M. biceps femoris, M. tibialis anterior, M. gastrocnemius medialis, M. deltoideus anterior part, M. deltoideus posterior part, M. latissimus dorsi. Electrode placement will follow the SENIAM guidelines. The skin underlying the electrode will be shaved and cleaned with alcohol to improve electrode-skin contact and reduce impedance.
* Reflective markers will be placed on fixed points of the lower and upper limbs of the patient. Marker placement will follow the Plug-in Gait full body model (VICON). For this model, the investigator will have to measure the following things in advance: body length, body weight, leg length, knee width, ankle width, shoulder offset, elbow width, wrist width, hand thickness.

After these preparations, patients will start to walk on the self-paced treadmill of the GRAIL system. For safety only, patients will walk with the safety harness. Patients will first be habituated to walking on the self-paced treadmill for 8 minutes without any form of VR. Patients need this habituation trial in order to get used to the self-paced treadmill system. After these 8 minutes, the treadmill will be stopped and patients will be seated for a 5-minute rest period. During the rest period, patients will be asked to fill in two short questionnaires (the Simulator Sickness Questionnaire-1, the VAS scales).

GRAIL session: After the 5-minute rest period, patients will walk for another 3 times 8 minutes with the VR. Patients are now walking while looking at a virtual environment that is projected onto the projection screen of the GRAIL device (semi-immersive). The optic flow will be different during each 8-minute walk. Between each walk, patients will rest for 5 minutes and during each rest period, patients will be asked to fill in a short questionnaire (the Simulator Sickness Questionnaire-2,-3).

HMD session: After the 5-minute rest period, patients will walk for another 3 times 8 minutes with the VR. Patients are now walking while wearing the HMD 'Oculus Rift' and are being fully immersed in a virtual environment (fully-immersive). The optic flow will be different during each 8-minute walk. Between each walk, patients will rest for 5 minutes and during each rest period, patients will be asked to fill in the a short questionnaire (the Simulator Sickness Questionnaire-2,-3).

To end both sessions, participants will be asked to fill in 3 questionnaires (the Simulator Sickness Questionnaire-Post, the VAS scales and the Igroup Presence Questionnaire).

RANDOMIZATION

First, the type of session will be randomized with 2 possible options: GRAIL - HMD or HMD - GRAIL. Second, the optic flow speed manipulation (matched, slow, fast) within the session will be randomized. The order of the manipulation will be the same in both sessions. The first 8 minutes in each session will always be the one without VR. Thereafter, the optic flow speed will be manipulated. There are 6 possible options for the randomization of the optic flow speed manipulation: matched - slow - fast / matched - fast - slow / slow - fast - matched / slow - matched - fast / fast - slow - matched / fast - matched - slow. The randomizations will be done through block randomization in Microsoft Excel®.

STUDY ANALYSIS

This study will investigate (1) the effect of manipulating the optic flow speed and (2) the effect of the level of immersion (semi-immersive GRAIL system with full-immersive HMD).

The effect optic flow speed has on the spatiotemporal gait parameters, kinematics, kinetics and muscle activity will be compared with walking without VR. In a first stage, the data will be visualized using LO(W)ESS smoothing (locally weighted scatterplot smoothing) to explore the observed effects over time (per condition and outcome), allowing for flexibility using this quasi-nonparametric approach. Next, relevant values expressing onset, magnitude and duration of the effect will be extracted:

* Onset: time point(s) at which the minimal clinically important difference (MCID) is exceeded. In case MCID is unknown, a 10% threshold will be used
* Magnitude: magnitude of the maximum (or maxima) and time point(s) at which the maximum is reached
* Duration: time between the onset and the time point at which the MCID (or 10% threshold) is no longer exceeded

These values will be compared between conditions in a two-way repeated measures ANOVA (optic flow speed * device). If relevant (based on the exploratory analyses), additional in-depth statistics, such as functional data analysis, will be performed under the guidance of the Department of Statistics and Data Analysis of our university.

ELIGIBILITY:
Inclusion Criteria stroke patients:

* diagnosed with stroke (as defined by the World Health Organization)
* stroke onset ≥ 3 months
* ambulatory with an impaired gait pattern (FAC-score 2, 3 or 4)
* ability to walk on a treadmill for 4x8 minutes without bodyweight support
* adult (≥ 18 years)
* ability to signal pain, fear and discomfort
* ability to give informed consent

Exclusion Criteria stroke patients:

* other neurological deficits than stroke leading to impaired gait (e.g. Parkinson's disease, multiple sclerosis)
* comorbidities (e.g. COPD, severe osteoporosis, cardiovascular instability)
* visual and/or vestibular disorders that can interfere with the VR
* uncontrolled spasticity significantly interfering with the movement of the lower extremities (Modified Ashworth Scale > 2)
* acute medical illness
* communicative/cognitive problems leading to the inability to understand and carry out instructions
* severe unilateral spatial neglect

Inclusion Criteria healthy people:

* ≥ 18 years of age
* normal or corrected-to-normal vision with glasses or contact lenses,
* no locomotion impairments

Exclusion Criteria healthy people:

* having a significant lower extremity injury during the last two years that might affect their gait
* having any type of vestibular/visual deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
3D kinematic measurements lower limb | through study completion, an average of 1 year
  Kinematic data (i.e. movement amplitudes of the bilateral hip, knee and ankle joint in degrees) of the lower limbs during treadmill walking will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
3D kinematic measurements upper limb (arm swing) | through study completion, an average of 1 year
  Kinematic data (i.e. movement amplitudes of the bilateral shoulder, elbow and wrist joint in degrees) of the upper limb during treadmill walking will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz. With these data, information about the arm swing during walking will be obtained.
3D kinetic measurements lower limb | through study completion, an average of 1 year
  Kinetic data (i.e. forces, moments and powers of the bilateral hip, knee and ankle joint in respectively Newton, Newton-meters and Watt) of the lower limbs during treadmill walking will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Walking speed | through study completion, an average of 1 year
  Walking speed (m/s) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Cadence | through study completion, an average of 1 year
  Cadence (steps/min) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Step length | through study completion, an average of 1 year
  Step length (cm) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Step time | through study completion, an average of 1 year
  Step time (s) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Swing - and stance time | through study completion, an average of 1 year
  Swing and stance time (s) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Single - and double limb support period | through study completion, an average of 1 year
  Single and double limb support period (% gait cycle) will be recorded continuously with the use of a 10-camera VICON Vero 1.3 system at 100 Hz.
Lower limb muscles activity | through study completion, an average of 1 year
  Muscle activity of the lower limb muscles (bilateral: M. rectus femoris, M. vastus lateralis, M. biceps femoris, M. tibialis anterior, M. gastrocnemius medialis) will be recorded continuously during treadmill walking with the use of surface electrodes. Signals will be recorded with the wireless EMG system Delsys Tigno (16 channels).
Upper limb muscles activity | through study completion, an average of 1 year
  Muscle activity of the upper limb muscles (bilateral: M. deltoideus anterior part, M. deltoideus posterior part, M. latissimus dorsi) will be recorded continuously during treadmill walking with the use of surface electrodes. Signals will be recorded with the wireless EMG system Delsys Tigno (16 channels).

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire | through study completion, an average of 1 year
  The Simulator Sickness Questionnaire (SSQ) is a widely used questionnaire to evaluate motion sickness when using VR. The SSQ consist of 16 symptoms divided in three components: nausea, oculomotor and disorientation. At the beginning of the session and after each 8 minute walk, participants need to indicate how much (none - slight - moderate - severe) each symptom is affecting them at that moment. The total score of the SSQ ranges between 0-235.62 points and higher scores indicate higher levels of simulator sickness.
Igroup Presence Questionnaire | through study completion, an average of 1 year
  The Igroup Presence Questionnaire (IPQ) is a scale for measuring the sense of presence experienced in a virtual environment. The IPQ consists of 14 questions divided in three subscales (spatial presence, involvement, experienced realism) and one additional general item not belonging to a subscale. The IPQ is scored on a 7-point Likert scale. After each session, participants will be asked to fill in the IPQ. The total score of the IPQ ranges between 0-98 points and higher scores indicate a higher sense of presence experienced in a virtual environment.
Visual Analogue Scale | through study completion, an average of 1 year
  After walking without the VR and after walking with the VR, participants will have to fill in two Visual Analogue Scales (VAS). Participants will have to indicate on a 100mm line how much they liked walking on the treadmill under these conditions (VAS1) and whether they would like to do this type of gait training during their rehabilitation (VAS2). The total score of the VAS scales ranges between 0-100 points and higher scores mean a better outcome.
Number of falls or stumbles | through study completion, an average of 1 year
  The number of falls or stumbles that patients experience will be noted in a standardized way.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, Prof. Ph.D, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Emma De Keersmaecker, Brussels, Belgium

REFERENCES:
- [Derived] De Keersmaecker E, Van Bladel A, Zaccardi S, Lefeber N, Rodriguez-Guerrero C, Kerckhofs E, Jansen B, Swinnen E. Virtual reality-enhanced walking in people post-stroke: effect of optic flow speed and level of immersion on the gait biomechanics. J Neuroeng Rehabil. 2023 Sep 25;20(1):124. doi: 10.1186/s12984-023-01254-0. PMID 37749566